CLINICAL TRIAL: NCT07392463
Title: Comparative Effects of Artificial Intelligence Teaching and Immersive Virtual Reality Smart Classroom Teaching on Children and Adolescents With ADHD: A Randomized Controlled Trial
Brief Title: Artificial Intelligence Versus Virtual Reality Teaching for Children and Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province (Other)
Responsible Party: Principal Investigator, Ning Li, Principal Investigator, Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THKX-ADHD-AI-VR-2024
Record Dates: First submitted 2026-01-25; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Artificial Intelligence; Virtual Reality; Digital Education; Executive Function; Children and Adolescents; Randomized Controlled Trial; Non-Pharmacological Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to either an artificial intelligence-assisted teaching group or an immersive virtual reality-based teaching group and received the assigned intervention in parallel throughout the study period.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the digital teaching interventions, participants and intervention providers were not blinded to group assignment. Outcome assessors were blinded to treatment allocation throughout data collection and evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Assisted Teaching Group (Experimental): Participants assigned to this arm received artificial intelligence-assisted teaching delivered through a tablet-based adaptive learning system. The intervention was conducted for 12 weeks, with three sessions per week and each session lasting approximately 45 minutes. The system incorporated real-time feedback and adaptive task adjustment based on individual learning performance and attention patterns.
  Interventions: Behavioral: Artificial Intelligence-Assisted Teaching
- Virtual Reality Smart Classroom Group (Experimental): Participants assigned to this arm received immersive virtual reality-based smart classroom teaching. The intervention was delivered using VR technology to simulate interactive learning scenarios in a low-distraction environment. The program was conducted for 12 weeks, with three sessions per week and each session lasting approximately 45 minutes.
  Interventions: Behavioral: Virtual Reality-Based Smart Classroom Teaching

INTERVENTIONS:
Behavioral: Artificial Intelligence-Assisted Teaching — A behavioral digital teaching intervention delivered through an artificial intelligence-assisted adaptive learning system. The system dynamically adjusted task difficulty and learning pace based on individual performance and attention-related behavioral data and provided real-time feedback during learning activities. The intervention was administered for 12 weeks, three sessions per week, with each session lasting approximately 45 minutes.
  Arms: AI-Assisted Teaching Group
Behavioral: Virtual Reality-Based Smart Classroom Teaching — A behavioral teaching intervention delivered using immersive virtual reality technology to simulate interactive classroom and task-based learning scenarios. Participants engaged in structured learning activities within a low-distraction virtual environment designed to enhance attention and engagement. The intervention was conducted for 12 weeks, three sessions per week, with each session lasting approximately 45 minutes.
  Arms: Virtual Reality Smart Classroom Group

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a common neurodevelopmental condition in children and adolescents and is often associated with difficulties in attention, behavior regulation, and executive functioning. In addition to medication, non-pharmacological interventions, including digital and technology-assisted educational approaches, have gained increasing interest.

This randomized controlled trial compared the effects of artificial intelligence (AI)-assisted teaching and immersive virtual reality (VR)-based smart classroom teaching on core ADHD symptoms and executive function in children and adolescents with ADHD. A total of 90 participants aged 8 to 15 years who met diagnostic criteria for ADHD were randomly assigned to either an AI-assisted teaching group or a VR-based teaching group.

Both groups received structured teaching interventions for 12 weeks, three sessions per week, with each session lasting 45 minutes. ADHD symptoms and executive function were assessed before the intervention, at the end of the intervention, and at a 3-month follow-up using validated rating scales.

The purpose of this study was to evaluate and compare the effectiveness of these two digital teaching approaches and to provide evidence for personalized, non-pharmacological educational interventions for children and adolescents with ADHD.

DETAILED DESCRIPTION:
This study was an open-label, randomized, parallel-group controlled trial designed to compare the effects of artificial intelligence (AI)-assisted teaching and immersive virtual reality (VR)-based smart classroom teaching on core symptoms and executive function in children and adolescents with attention-deficit/hyperactivity disorder (ADHD).

Participants aged 8 to 15 years were recruited from an outpatient ADHD clinic and were required to meet diagnostic criteria for ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Eligible participants were randomly assigned in a 1:1 ratio to either the AI-assisted teaching group or the VR-based teaching group using a computer-generated randomization sequence prepared by an independent statistician. Due to the nature of the digital interventions, participants were not blinded to group allocation; however, outcome assessments were conducted by trained evaluators who were blinded to treatment assignment.

Both groups received structured teaching interventions for 12 weeks, with three sessions per week and each session lasting approximately 45 minutes. The AI-assisted teaching intervention was delivered using a tablet-based adaptive learning system incorporating eye-tracking, behavioral analysis, and real-time feedback to dynamically adjust task difficulty and learning pace based on individual performance and attention patterns. The VR-based teaching intervention was delivered using immersive virtual reality technology to simulate classroom and task-based learning scenarios, with an emphasis on interactive learning and emotional regulation in a low-distraction environment.

Primary outcomes included changes in core ADHD symptoms as measured by the ADHD Rating Scale (ADHD-RS). Secondary outcomes included changes in executive function assessed using the Behavior Rating Inventory of Executive Function (BRIEF), parent-report version. Outcome measures were assessed at baseline prior to intervention initiation, at the end of the 12-week intervention period, and at a 3-month post-intervention follow-up.

All study procedures were approved by the Ethics Committee of Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, and written informed consent was obtained from parents or legal guardians, with assent obtained from participating children when appropriate. The study was conducted in accordance with the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 8 to 15 years.
* Diagnosis of attention-deficit/hyperactivity disorder (ADHD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), confirmed by two qualified child psychiatrists.
* Total score of 25 or higher on the ADHD Rating Scale (ADHD-RS).
* Intelligence quotient (IQ) of 80 or above as assessed by the Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV).
* Stable clinical status for at least 30 days prior to enrollment, with adherence to standard first-line or second-line treatment regimens, and no planned changes in treatment during the study period.
* Ability to participate in structured digital teaching sessions.
* Written informed consent provided by a parent or legal guardian, with assent obtained from the participant when appropriate.

Exclusion Criteria:

* Presence of neurodevelopmental or neurological disorders other than ADHD, such as cerebral palsy or epilepsy.
* Diagnosis of severe psychiatric disorders, including schizophrenia.
* Significant sensory impairments (e.g., hearing impairment) that could interfere with study participation.
* Lack of response to two or more different classes of ADHD medications.
* History of suspected substance abuse or dependence within the past 6 months.
* Physical conditions or motor impairments that would prevent participation in the teaching interventions.
* Current suicidal ideation or severe suicidal behavior as determined by the investigator.
* Receipt of other structured psychological or educational interventions during the study period.
* Any other condition that, in the opinion of the investigator, would make participation in the study inappropriate.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Core ADHD Symptoms Measured by the ADHD Rating Scale (ADHD-RS) | Baseline and at the end of the 12-week intervention period
  Core symptoms of attention-deficit/hyperactivity disorder (ADHD) were assessed using the ADHD Rating Scale (ADHD-RS), which includes subscales for inattention and hyperactivity/impulsivity. Higher scores indicate greater symptom severity. The scale was completed by trained evaluators based on standardized assessment procedures.

SECONDARY OUTCOMES:
Change in Executive Function Measured by the Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, at the end of the 12-week intervention period, and at the 3-month post-intervention follow-up
  Executive function was assessed using the parent-report version of the Behavior Rating Inventory of Executive Function (BRIEF), which evaluates multiple domains including inhibition, working memory, planning/organization, and emotional control. Higher scores indicate greater impairment in executive function.
Change in Inattention Symptoms Measured by the ADHD Rating Scale (ADHD-RS) Inattention Subscale | Baseline, at the end of the 12-week intervention period, and at the 3-month post-intervention follow-up
  Inattention symptoms were assessed using the inattention subscale of the ADHD Rating Scale (ADHD-RS). The subscale consists of items evaluating attention-related difficulties, with higher scores indicating more severe inattention symptoms.
Change in Hyperactivity/Impulsivity Symptoms Measured by the ADHD Rating Scale (ADHD-RS) Hyperactivity/Impulsivity Subscale | Baseline, at the end of the 12-week intervention period, and at the 3-month post-intervention follow-up
  Hyperactivity and impulsivity symptoms were assessed using the hyperactivity/impulsivity subscale of the ADHD Rating Scale (ADHD-RS). Higher scores reflect greater severity of hyperactivity and impulsivity symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, PhD, Principal Investigator — Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province
Locations (1):
- Hongxinkang New Traditional Chinese Medicine Hospital, Tongren, Tongren, Guizhou, China

IPD SHARING:
Plan to Share IPD: No